CLINICAL TRIAL: NCT05214014
Title: Treatment of Patients With Systemic Sclerosis With Autologous Regulatory Т-cells
Brief Title: Treatment of Systemic Sclerosis With Autologous Regulatory Т-cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_TREGS
Record Dates: First submitted 2021-11-29; First posted 2022-01-28 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with systemic sclerosis receiving standard treatment and autologous regulatory Т-cells (Experimental): Group 1: Patients with systemic sclerosis receiving standard treatment and autologous regulatory Т-cells
  Interventions: Biological: Autologous Regulatory Т-cells; Other: Standard treatment according to the clinical protocols
- Patients with multiple sclerosis receiving standard treatment (Active Comparator): Group 2: Patients with multiple sclerosis receiving standard treatment
  Interventions: Other: Standard treatment according to the clinical protocols

INTERVENTIONS:
Biological: Autologous Regulatory Т-cells — Autologous Regulatory Т-cells obtained from CD4+CD25+ cells isolated from PBMC and cultured with the cocktail of cytokines and antibodies to induce proliferation of Tregs
  Arms: Patients with systemic sclerosis receiving standard treatment and autologous regulatory Т-cells
Other: Standard treatment according to the clinical protocols — Standard treatment of Systemic Sclerosis according to the clinical protocols

SUMMARY:
Treatment of patients with systemic sclerosis with autologous regulatory Т-cells

DETAILED DESCRIPTION:
Considering the fact that a decrease in the content and functional activity of T-reg plays an important role in the immunopathogenesis of many systemic diseases of the connective tissue, the use of a large amount of T-reg can have a therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Systemic Sclerosis
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* The presence of any malignant tumor within the last 5 years
* Acute or chronic diseases in the stage of decompensation
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding, or fertile patients who are not using adequate contraceptive methods
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ACR/EULAR systemic sclerosis criteria | 6 month
  Сalculation of ACR/EULAR systemic sclerosis criteria score
ACR/EULAR systemic sclerosis criteria | 1 year
  Сalculation of ACR/EULAR systemic sclerosis criteria score
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Kanstantsin Chyzh, Dr, Study Director — Belarusian State Medical University
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No